CLINICAL TRIAL: NCT04543669
Title: Adacel® (TdaP-Tetanus, Diphtheria, Acellular Pertussis) Booster Vaccination of Acellular Pertussis Vaccine-primed Individuals for Cell Mediated Immunity Assay Development
Brief Title: Adacel® Booster Vaccination for CMI Assay Development
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry); VaxDesign Corporation (Unknown)
Responsible Party: Principal Investigator, Scott Halperin, Professor and Director, Canadian Centre for Vaccinology, Dalhousie University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SP1601
Record Dates: First submitted 2017-04-26; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Pertussis
MeSH Terms: conditions — Whooping Cough | interventions — adacel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Adacel® (Experimental): All participants will receive one booster dose of commercially available Adacel® (TdaP-Tetanus, diphtheria, acellular pertussis) vaccine
  Interventions: Biological: Adacel®

INTERVENTIONS:
Biological: Adacel® — Vaccine for TdaP-Tetanus, diphtheria, acellular pertussis

SUMMARY:
Recruitment of individuals primed during childhood with TdaP (tetanus, diphtheria , acellular pertussis) vaccine, and administration of an Adacel booster with blood sample collection at various time points before and after vaccination.

Collection of blood sample volumes will be large enough to allow assessment and comparison of multiple assays that evaluate cell-mediated immune (CMI) responses and other biomarkers following the administration of pertussis vaccinations. The ultimate objective would be to utilize these validated assays for evaluation of pertussis clinical trial results or development of new pertussis vaccine formulations.

DETAILED DESCRIPTION:
Pertussis, known as "whooping cough", is caused by the bacterium Bordetella pertussis which was discovered over a century ago. Human vaccines were developed in the subsequent two decades and routine childhood immunization has been practiced for over 60 years. Yet, B. pertussis remains a significant cause of morbidity in children and adults worldwide. Globally, about 20-40 million cases of pertussis are reported each year, with about 400,000 cases being fatal. The incidence of pertussis is highest and the severity the greatest in children under 6 months of age. Vaccination and natural infection are not protective for life, and the reason is unclear. The epidemiologic features of B. pertussis infections in older individuals who are only partially immune from prior infections and immunizations are not well understood. Clarification is important, in light of studies that suggest that pertussis is a cause of prolonged cough illness in adults who serve as the reservoir of B. pertussis and are the major source of infection for infants in whom the disease has substantial morbidity and mortality. With the considerable increase in cases and outbreaks, there is an imminent need for improved immunogenic and efficacious pertussis vaccines, paired with the best tools to evaluate vaccines and vaccine programs.

VaxDesign has proposed two studies for acellular vaccine primed (acP) versus whole cell vaccine primed (wcP) donors, to further develop and validate a number of practical assays for use as biomarkers and to define a baseline readout for pertussis vaccinations from these two cohorts. In addition, these assays will be optimized to use the small blood volumes that are routinely available from clinical studies. In contrast to measuring humoral immune responses, the cell mediated immune response (CMI) is a substantially more challenging parameter to assess and thus the sample volumes required for the study must be large enough to allow the multiple different assessments. In this study, samples will be taken to evaluate transcriptomics, and humoral and cellular immunity over a one month period following vaccination. The collaboration with the Canadian Center for Vaccinology (CCfV) offers a unique opportunity of easily accessing acellular vaccine primed individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16years
* Primed during infancy with an acellular pertussis vaccine
* Good general health status, as determined by history no greater than 30 days prior to administration of the first test article
* Written informed consent provided
* If female of child-bearing potential, has a negative pregnancy test on the day of consent and has agreed to continue adequate contraception until after the last blood draw.

Exclusion Criteria:

* Not primed in infancy with an acellular pertussis vaccine
* History of anemia
* Underlying chronic medical condition requiring ongoing monitoring by a physician (e.g., diabetes, seizure disorder)
* Underlying cardiac and/or pulmonary disease including hypertension, angina, prior myocardial infection, asthma, emphysema, chronic bronchitis, and pulmonary tuberculosis
* Pregnant (known before or established at the time of screening using a urine-based test)
* Immunocompromised (reporting HIV/AIDS positive or receiving immunosuppressive therapy involving steroids)
* Vaccinated against pertussis within previous 5 years
* Refusing to get an Adacel® (TdaP) vaccination dose

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Determine best assay to evaluate CMI responses post-vaccination: CD4 T-cell proliferation | Days -14 to 28
  % CD4+CTV-T cells analyzed by flow cytometry
Determine best assay to evaluate CMI responses post-vaccination: CD8 T-cell proliferation | Days -14 to 28
  % CD8+ CTV-T cells analyzed by flow cytometry
Determine optimal time point for sample collection: CD4 T-cell responses | Days -14 to 28
  % CD4+CTV-cytokine+T cells analyzed by flow cytometry
Determine optimal time point for sample collection: CD8 T-cell responses | Days -14 to 28
  % CD8+ CTV-cytokine+T cells analyzed by flow cytometry

SECONDARY OUTCOMES:
Transcriptomic profiling of host - B. pertussis antigen interactions: B-cell plasmablasts | Days -7, 7, 14, and 28
  ASC per 106 PBMCs (ELISpot)
Transcriptomic profiling of host - B. pertussis antigen interactions: B-cell plasmablasts | Days -7, 7, 14, and 28
  % CD19+ CD38+ CD27+ cells

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Halperin, MD, Principal Investigator — Dalhousie
Locations (1):
- Canadian Center for Vaccinology, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No